CLINICAL TRIAL: NCT03491345
Title: A Phase II Study of Avelumab Monotherapy in PD-L1 Positive or EBV Positive or MSI-H or POLE/POLD1 Mutated Advanced Solid Tumor (Part of K-BASKET Trial; Korea-Biomarker-driven Multi-arm Drug-screening, Knowledge and Evidence-generating Targeted Trial)
Brief Title: K-Basket, Avelumab, Biomarker-driven, Advanced Solid Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-1142
Record Dates: First submitted 2018-03-30; First posted 2018-04-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: PD-L1 Positive Mutation Tumor; EBV Positive Mutation Tumor; MSI-H Mutation Tumor; POLE/POLD1 Mutation Tumor
MeSH Terms: interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- avelumab (Experimental)
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — avelumab 10mg/kg, IV, q 2 weeks

SUMMARY:
Investigators have conducted K-BASKET trial (Korea-Biomarker-driven multi-arm drug-screening, knowledge and evidence-generating targeted trial), which was based on the specific genetic aberration, not the cancer type, which could accelerate matching the right drug to the right target so that every cancer patient could get the right specific drug based on the specific genetic biomarker, like NCI-MATCH trial. Next generation sequencing (NGS) focusing panel has the mutation and copy number variation of MET, PIK3CA and AKT. Investigators will open new treatment arms during the progress of K-BASKET trial. Patient with PD-L1 positive or EBV positive or MSI-H or POLE/POLD1 mutation tumor will be assigned to Avelumab monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent for treatment.
* Age ≥ 20 years old
* Meet at least one of the following requirements; A. PD-L1 positive by IHC or B. EBV positive by ISH or C. MSI-H by IHC or D. POLE mutation E. POLD1 mutation
* Progressive disease who failed to previous standard treatment
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 on time of patient's allocation.
* Adequate organ function as defined by the following criteria:

A. Adequate hematological function defined by absolute neutrophil count (ANC) ≥ 1500/mm3, platelet count ≥ 100,000/mm3 , hemoglobin ≥ 9.0 g/dL B. Adequate hepatic function defined by AST and ALT levels ≤ 2.5 × upper limit of normal (ULN) and total bilirubin level ≤ 1.5 × ULN C. Adequate renal function defined by and estimated creatinine clearance (CrCl) ≥ 30 mL/min (MDRD)

* A life expectancy of at least 90 days
* Negative serum pregnancy test at screening for women of childbearing potential
* Highly effective contraception for both male and female subjects if the risk of conception exists.

Exclusion Criteria:

* Previous treatment with immune checkpoint inhibitor (Anti-PD1, Anti-PDL1, Anti-CTLA4 etc.)
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI CTCAE v 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
* Prior organ transplantation, including allogeneic stem cell transplantation
* Significant acute or chronic infections
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:
* All subjects with brain metastases, except those meeting the following criteria:
* Subjects with clinically significant (i.e., active) cardiovascular medical history: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
* Unresolved toxicity of Grade >1 attributed to any prior therapies (excluding alopecia, skin pigmentation and anemia).
* Pregnancy or lactation
* Interstitial lung disease
* Known alcohol or drug abuse
* All other significant diseases (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 6 weeks

SECONDARY OUTCOMES:
safety assessed by CTCAE v4.0 | 2 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
disease control rate | 6 weeks
progression free survival | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Medical Oncology, Severance Breast Cancer Clinic, Yonsei Cancer Center, Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided